CLINICAL TRIAL: NCT07099300
Title: The Use of Nasogastric Tubes and Water-Soluble Contrast With or Without Radiographic Imaging in The Management of Adhesive Small Bowel Obstruction: A Feasibility Study
Brief Title: Water-Soluble Contrast Induced Intestinal Stimulation for the Treatment of Small Bowel Obstruction: A Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edward Harry Livingston, Professor of Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-6143
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Small Bowel Obstruction
Keywords: water soluble contrast; radiology
MeSH Terms: interventions — Radiography, Abdominal

STUDY DESIGN:
Intervention Model Description: Parallel Group, Randomized, Clinical Trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging (Experimental): Patients with SBO will undergo an initial WSC study but no subsequent x-rays will be obtained,
  Interventions: Diagnostic Test: Abdominal Radiography
- Control (Active Comparator): Patients with SBO will undergo an initial WSC study and will have routine abdominal radiographs at 12, 24, and 48 hours.
  Interventions: Diagnostic Test: Abdominal Radiography

INTERVENTIONS:
Diagnostic Test: Abdominal Radiography — Obtain plain film radiographs 3 times after adminstration of WSC

SUMMARY:
Small bowel obstruction (SBO) is common yet, how to best manage it remains unknown. One approach is to administer water soluble oral contrast (WSC) and the obtain x-rays to determine how well the bowel is functioning. WSC may help resolve SBO by stimulating the bowel by itself. The intent of this study is to determine if the x-ray component of this therapeutic approach is necessary.

DETAILED DESCRIPTION:
Responsible for more than 340,000 hospital admissions per year, small bowel obstruction (SBO) is one of the most common causes of serious gastrointestinal disease in the US. Adhesion-related SBO (aSBO) is usually treated by the placement of a nasogastric tube (NGT) to decompress the stomach, administration of intravenous (IV) fluids and observation by a surgical team. In most (60%) patients, aSBO resolves spontaneously. However, NGTs are uncomfortable for patients and have multiple associated risks, leading many patients and clinicians to avoid their use if possible.

Despite NGT placement being considered a standard component of aSBO treatment, some series report that as many as ½ of all patients with aSBO may be treated without them. A recent meta-analysis showed that hospital length-of-stay (HLOS) may be reduced by 2 days if treated with water-soluble contrast (WSC).

Despite aSBO being common, little is known about the optimal means for its treatment and even less about the mechanisms by which it resolves. The overall intent of this research is to develop evidence-based treatment protocols and to better understand the mechanisms by which aSBO resolves and how interventions can be developed to improve its treatment.

This feasibility study's purpose is to determine the ability to perform a randomized clinical trial (RCT) investigating treatments options for aSBO. Specifically, WSC will be administered to patients with a SBO followed by randomization to undergo formal upper gastrointestinal-small bowel follow through (UGI-SBFT) series vs no radiologic imaging to determine if radiologic examination can be eliminated when treating patients with aSBO. A concurrent observational arm will enroll patients who elect not to have NGTs placed to follow their hospital course. A state-transition model of daily clinical status will be tested to determine its effectiveness as a primary outcome to replace older, traditional outcomes for hospitalized patients such as diet resumption or length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of aSBO as evidenced by one or more clinical features meeting the following criteria:

   * Nausea
   * Emesis
   * Abdominal pain
   * Distended abdomen
   * CT evidence of aSBO
   * Known abdominal surgical history.
2. Written informed consent obtained from subject.

Exclusion Criteria:

1. Unable to provide consent for the study.
2. Pregnant or breastfeeding.
3. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
4. Unstable angina or recent myocardial infarction or stroke within 6 months
5. Patients with peritonitis or who require immediate surgery.
6. Non-adhesive SBO, including.

   * Paralytic Ileus
   * Incarcerated hernia
   * Fecal impaction
   * Intra-abdominal malignancy
   * Early aSBO within 4 weeks of a prior abdominal operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2030-08-15 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Median number of days of benefit | 30 Days
  probability distribution of the difference in median number of days of benefit attributable to the intervention determined from the posterior distribution of state occupancy probabilities.

SECONDARY OUTCOMES:
Daily Clinical Status | 30 day
  longitudinal, ordinal state transition analysis of a patient's clinical status on any day within a 30-day window
Health Care Quality of Life (HCQOL) | 30 Day
  HCQOL as assessed by PROMIS-29: Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) has a physical function scale ranging from 30-56 with higher scores representing better physical function. Anxiety, depression, fatigue, sleep disturbance, social function, pain interference have scales ranging from a low of 30-40 and a high of 60-80 with higher scores representing worse outcomes. Pain intensity is measured on a scale of 0 to 10 with 10 representing more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Edward H Livingston, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No
The study will be of patients who are potentially identifiable. Data will not be publically available to protect their identities.